CLINICAL TRIAL: NCT00687518
Title: Effects of Intravenous Injection of Erythropoietin on Hepcidin Pharmacokinetics in Healthy Volunteers
Acronym: HEPEPO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Direction of Clinical Research and Strategy, Rennes University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DGS 2006/0416; CIC0203/056
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2008-05

CONDITIONS: Iron Metabolism Disorders
MeSH Terms: conditions — Iron Metabolism Disorders | interventions — Erythropoietin; epoetin beta

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): erythropoietin
  Interventions: Drug: Erythropoietin
- 2 (Placebo Comparator): Saline serum
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erythropoietin — Intravenous injection of 50 U/kg of erythropoietin
  Other Names: Neorecormon®
  Arms: 1
Drug: Placebo — Intravenous injection of equivalent volume of saline serum
  Other Names: NaCl 0,9%
  Arms: 2

SUMMARY:
The aim of this study is to measure the variations of serum and urinary hepcidin levels following a single intravenous injection of erythropoietin in healthy volunteers. Hepcidin is a major regulator of iron homeostasis. It acts by binding on ferroportin, and limits cellular efflux of iron through enterocytes and macrophages. Anemia and hypoxia are known to modulate hepcidin synthesis. In these situations, erythropoietin synthesis is increased, so it can be postulated that erythropoietin could modulate hepcidin synthesis.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* male aged 18 - 30
* normal routine laboratory values
* normal ECG
* normal iron status

Exclusion Criteria:

* C282Y mutation of the HFE gene
* alcohol or tobacco consumption

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-11 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
serum hepcidin levels | over 24 hours

SECONDARY OUTCOMES:
urinary hepcidin levels | over 24 hours
serum iron and ferritin levels | over 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice LAINE, MD, Principal Investigator — Rennes University Hospital; Bruno LAVIOLLE, MD, Study Chair — RennesUniversity Hospital
Locations (1):
- Unité d'Investigation Clinique - Centre d'Investigation Clinique - Hôpital de Pontchaillou, Rennes, France

REFERENCES:
- [Derived] Laine F, Laviolle B, Ropert M, Bouguen G, Morcet J, Hamon C, Massart C, Westermann M, Deugnier Y, Loreal O. Early effects of erythropoietin on serum hepcidin and serum iron bioavailability in healthy volunteers. Eur J Appl Physiol. 2012 Apr;112(4):1391-7. doi: 10.1007/s00421-011-2097-7. Epub 2011 Aug 5. PMID 21818622